CLINICAL TRIAL: NCT04222335
Title: Understanding and Overcoming the Early Adaptive Resistance to EGFR Tyrosine-kinase Inhibitors in Lung Cancer Patients
Acronym: LUNG-RESIST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/18/0475; Numéro ID RCB : 2019-A02440-57 (Other: ANSM)
Record Dates: First submitted 2019-12-17; First posted 2020-01-09 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Lung Cancer, Nonsmall Cell
Keywords: Lung cancer; Targeted therapy; resistance
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood sampling (Other): Blood sampling
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — Each participant will be followed-up regularly as part of the usual practice for imaging and medical consultations. During their visits, from inclusion (T0) to the end of study participation (T progression), each patient will have a blood sampling specifically for the research to analyze tumor DNA and circulating tumor cells: T0, T1month, T3 months, Tn months, T DNA C+, T progression.
  This research does not include any other act or intervention specifically required for its purposes.

SUMMARY:
Epidermal growth factor receptor-tyrosine kinase inhibitors (EGFR-TKI) are effective therapies for advanced lung cancer patients bearing EGFR-activating mutations, but are not curative due to the invariable apparition of resistances. The investigator team have identified a new phenotype related to drug tolerance after EGFR-TKI treatment that shares several characteristics of a known process of Therapy-Induced Senescence (TIS), which could be a major event of drug tolerance in patients. Using cutting-edge technologies, patient-derived xenografts (PDX) and circulating tumor cells (CTC), the investigator team will perform an exhaustive characterization of the phenotypic and molecular changes associated with this drug-tolerant state in patients. Their results should lead to new therapeutic approaches to eliminate the reservoir of drug-tolerant cells and to prevent emergence of resistance mutations responsible for the relapse of patients.

DETAILED DESCRIPTION:
LUNG-RESIST is a translational, monocentric and prospective research study on 40 patients whose objective is to characterize Drug Tolerant Cell (DTC) type cells in patients with a NSCLC carrying an EGFR mutation and to discover and monitor potentials biomarkers involved in this mechanism of resistance to osimertinib. The study will be offered to patients, and for whom the therapeutic decision was decided collegially during multidisciplinary molecular meetings (molecular Tumor Board). Following informed consent, patients will be registered in a single cohort. In this study, treatment with osimertinib is not studied and will be delivered according to current recommendations

ELIGIBILITY:
Inclusion Criteria:

* Patient with non operable and / or metastatic non-small cell lung cancer documented histologically.
* Pathological diagnosis of NSCLC carrying an EGFR activating mutation associated with sensitivity to the tyrosine kinase inhibitors (TKI) (exons 18, 19 and 21).
* Sufficient tissue sample quantity and quality for translational research
* Naïve TKI-treated EGFR patient who can receive first-line treatment with Osimertinib or second-line after chemotherapy

Exclusion Criteria:

* Any patient with an exon 20 EGFR mutation.
* Any disease or pathology that recommend not to perform blood samples collection
* Any psychological, family, geographical or social condition that could potentially, according to the investigator's judgment, prevent the collection of informed consent or interfere with compliance with the study protocol
* Patient with a resistance mutation of EGFR
* Patient under State Medical Assistance
* Patient deprived of liberty on administrative or judicial decision, or patient under guardianship, curatorship or safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-03-26 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Rate of EGFR mutated patients for whom phenotypic characterization of DTC-like and osimertinib-tolerant tumor cells is feasible. | Up to one year or progression
  Rate of EGFR mutated patients for whom the DTC phenotype has been characterized at T0 (Baseline), T1 month, T3 month, Tn month, T antideoxyribonuclease (ADN) Circulant+, T progression

SECONDARY OUTCOMES:
Rate of patients for whom the molecular characterization of DTC-like cells is successfully performed. | Up to one year or progression
  This rate id defined by the number of patients who are successful compared to the total number of patients. Failure is defined by a patient with circulating tumor cells for which molecular characterization of DTC-like cells could not be performed at all measurement times.
Progression-free survival (PFS) | Up to one year or progression or death
  PFS is defined as the delay between the date of the patient's inclusion and the date of progression or death. Patients alive and without progression will be censored on the date of last news or on the date of initiation of a new anti-cancer therapy (if applicable).

CONTACTS AND LOCATIONS:
Overall Officials: Julien MAZIERES, MD; PHD, Principal Investigator — Toulouse University Hospitals
Locations (1):
- Toulouse University Hospital, Toulouse, Occitanie, France

IPD SHARING:
Plan to Share IPD: No